CLINICAL TRIAL: NCT06812156
Title: Evaluation of the Effectiveness of Nursing Interventions Aimed at Improving Cardiovascular Health Behaviors in Children
Brief Title: Cardiovascular Health and Nursing Interventions in 6th Grade Middle School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ozge Surel, nurse, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AnkaraN
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases (CVD); Cardiovascular Diseases Risk; Health Behavior; School Health Services; Nursing Care; Virtual Reality; Students of the 6. Grade; Nursing Education
Keywords: Child; Cardiovascular Diseases; Health Behavior; School Health; Nursing Intervention; Virtual Reality
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: The intervention study model involves a controlled and intervention-based approach to evaluate the impact of a variable in a specific population. In the study, educational and awareness-raising activities, as well as augmented reality technologies, were implemented in the intervention groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Other): A group of 43 sixth-grade students in the experimental group received five sessions of education on cardiovascular health, followed by a virtual reality video viewing session using VR goggles.
- control group (No Intervention): The 47 students in the control group did not receive any intervention; only measurements were conducted.

INTERVENTIONS:
Other: Cardiovascular Health Education — This intervention aims to promote healthy behavioral changes at both individual and community levels by supporting education with virtual reality technology.

SUMMARY:
Interventions that can improve cardiovascular health behaviors in children are of critical importance for reducing the burden of cardiovascular disease in the future. The research will be conducted to evaluate the effectiveness of nursing interventions aimed at improving heart health in children. The study employs a pre-test post-test control group experimental design. The sample of the study consists of a total of 100 students, with 50 in the experimental group and 50 in the control group. The research will be conducted with students from two middle schools selected through simple random sampling method from Mamak district, Ankara province. Socio-demographic Data Collection Form and Cardiovascular Health Behavior Scale for Children will be used during the data collection process. A 5-week educational plan aimed at improving cardiovascular health behaviors will be implemented for the experimental group, while no intervention will be made for the control group. Research data will be analyzed using Statistical Package for Social Sciences (SPSS) 25.0 program. Continuous variables will be reported using mean (x̅) and standard deviation (SD), while number (n) and percentage (%) will be used for categorical variables.

All tests will consider statistical significance at the level of p < 0.05. For the study to be conducted, ethical approval will be obtained from the Ankara University Rectorate Ethics Committee, institutional permission will be obtained from the Ankara Provincial Directorate of National Education, and verbal consent from the included students and written consent from their parents will be obtained.

DETAILED DESCRIPTION:
The school-age period is a phase where healthy behaviors can naturally be adopted and sustained throughout life. Unhealthy habits acquired during childhood are highly likely to lead to unhealthy adults (Arnaiz et al., 2021). Early age can be a key period for interventions, and the younger the intervention age, the more positive the outcomes. Therefore, a comprehensive healthy lifestyle intervention is needed in school settings as early as possible to reduce future cardiovascular disease risks (Dong et al., 2021). School-based initiatives are crucial in primary prevention programs for cardiovascular diseases (Yu et al., 2022). School-based programs for preventing cardiovascular diseases significantly contribute to the prevention of cardiovascular risk factors in children.Improving the content and practices of school-based cardiovascular disease prevention programs is essential to enhance their effectiveness. Integrating these programs into school curricula can significantly contribute to increasing their impact and widespread adoption (Amoah et al., 2021). It is necessary to promote ideal cardiovascular health in all children and improve the condition of those already experiencing cardiovascular health issues (Steinberger et al., 2016).

In a school-based study, interventions aimed at reducing cardiovascular risk factors were implemented, resulting in improvements in physical activity and fruit and vegetable consumption. Additionally, there was a decrease in the consumption of sugary foods and beverages as well as fried foods (Woodgate & Sigurdson, 2015). School-based cardiovascular health promotion initiatives contribute to increasing children's awareness of this issue. Strategies to foster a healthy lifestyle support cardiovascular health. Developing strategies to improve children's cardiovascular health is critical for reducing the burden of cardiovascular disease in the future (Woodgate & Sigurdson, 2015).

In a school-based obesity intervention study conducted in China, a reduction in the risk of overweight, obesity, and hypertension was observed in children aged 6-18 years. It was found that this reduction was greater in children aged 6-12 years compared to those aged 13-18 years (Dong et al., 2021).

According to the International Council of Nurses (2015), nurses, who represent the largest discipline in global healthcare, manage cardiovascular disease (CVD) risk factors and chronic diseases. The American Heart Association (AHA) and the World Health Organization (WHO) recognize the key role of nurses and other healthcare team members in supporting the goal of reducing CVD-related deaths and disabilities by 25% by 2025 (Smith et al., 2012; Yusuf et al., 2015). For over 40 years, nurses have played a crucial role in managing single and multiple risk factors through specialized clinics focused on hypertension, smoking, lipids, and diabetes, as well as through primary healthcare services, workplace programs, and cardiac rehabilitation initiatives (Miller & Froelicher, 2004; Fonarow et al., 2001).

Nurses have assumed a primary role as team leaders in providing case management, not only reducing CVD risk factors but also demonstrating their ability to adhere to treatment guidelines and protocols, reduce hospital admissions, and decrease morbidity and mortality in patients with heart disease (Berra et al., 2011; Berra, 2011; Allen et al., 2014). In the early 1990s, the SCRIP (Stanford Coronary Risk Intervention Project) study demonstrated that nurse-led risk reduction in patients with known CVD resulted in angiographically documented regression of the disease and a decrease in clinical events (Haskell et al., 1994). Following this landmark study, a series of clinical trials documented the significant and effective role of nurses in improving adherence to guideline-based medical treatments and lifestyle changes (Miller & Froelicher, 2004; Wood et al., 2008). The Cardiac Hospitalization Atherosclerosis Management Program showed a significant reduction in morbidity and mortality one year after discharge among patients who received nurse-led case management compared to those receiving usual care (Fonarow et al., 2001).The nursing profession plays a significant role in the prevention and control of cardiovascular diseases. School health nurses make substantial efforts to reduce the impact of cardiovascular diseases through responsibilities such as early diagnosis and intervention, education on healthy lifestyle changes, raising community awareness, monitoring risk factors, fostering family and community collaboration, and emergency management (Ministry of Health, 2015). It is essential for all nurses, particularly school health nurses, to have high levels of knowledge and awareness regarding cardiovascular diseases and their risk factors. Nurses should evaluate children they encounter in their work environments for cardiovascular disease risk factors, collect information from parents and children about these risk factors, and educate children and their families at high risk about the necessary precautions. Nurses should collaborate with schools to expand school-based cardiovascular health promotion initiatives and efforts to prevent cardiovascular disease risk factors (Hayman et al., 2015).

Virtual reality (VR) is defined as a multimedia technology that appeals to human senses to enhance the interaction between the real and virtual worlds (Stone, 1991; Oppenheim, 1993). It uses advanced technological devices to provide users with a sense of being surrounded by a virtual environment and experiencing a realistic simulation through immersive visuals and sounds (Skalicky & Kong, 2019; Binay & Bal, 2021). Virtual reality headsets are equipped with adjustable straps and a device on the front that allows users to feel as if they are in a different reality by simultaneously experiencing various senses. The ability of therapeutic virtual environments to create a sense of reality distinguishes VR headsets from other applications (Banos et al., 2013; İnan, 2017). Through 360-degree content design, VR headsets offer users a seamless exploration experience in the virtual world, regardless of the direction they look (Jokela et al., 2019).

Virtual reality is a technology that allows users to feel as if they are genuinely present in a computer-generated three-dimensional environment. Over the past two decades, it has been used for various purposes in the healthcare field (Indovina et al., 2018; Guerra-Armas et al., 2023; Musters, Vandevenne, Franx & Wassen, 2023). In a doctoral dissertation completed in 2020, Caner examined the effects of VR headsets and smartphone gaming applications on preoperative anxiety in children aged 7-13 years (Caner, 2020). In 2021, Turgut conducted a master's thesis study with hospitalized children aged 4-10 years and their parents. In this study, the control group received standard care, while the VR group watched a tour video with headsets before surgery and cartoons post-surgery. The results showed that VR headsets reduced anxiety and pain in children while increasing parental satisfaction (Turgut, 2021). In Kurban's 2022 master's thesis, it was determined that the use of VR headsets during vaccination in children aged 6-12 years was effective in reducing pain and anxiety levels (Kurban, 2022). In another doctoral dissertation, the effects of using virtual reality (VR) headsets during school vaccinations on children's fear and anxiety levels were examined, and it was found that the use of VR headsets was effective in managing fear and anxiety (Kırbaş, 2021).

Traditional teaching methods are increasingly inadequate in meeting the needs of students and teachers. Consequently, administrators and researchers are turning to technological tools to develop effective teaching models. One such tool is virtual reality technologies, which enhance student-teacher interaction (Şenol, 2018). VR technologies not only provide a rich teaching model in education but also help students develop new ideas and problem-solving skills. These technologies combine interactive, imaginative, and three-dimensional visualization techniques to offer students an entirely accessible virtual learning environment. This environment allows students to express, create, or do anything they desire at any time (Pan, Cheok, Yang, Zhu & Shi, 2006).

In Gedik's 6th-grade class, lessons on different climates around the world were supported with VR headsets. At the end of the lessons, a survey was conducted to determine the impact of VR technology on the classes. The results showed that VR technology increased students' interest in social studies and helped them better understand climate topics (Rüştü, 2020). Other studies have also supported this perspective (Başaran, 2010; Çoruh, 2011; Arıcı, 2013; Çağıltay et al., 2001; Demirli, 2000). Tanrıverdi's (2017) doctoral thesis investigated the effects of balance training in children and compared exercise game systems with conventional methods. The results suggested that exercise game systems could be an effective tool for improving balance skills in children (Tanrıverdi, 2017).

Another study examined the potential development of certain muscle strength parameters in children who participated in virtual reality sports applications for eight weeks. The findings revealed significant differences in movements such as left and right knee flexion, knee extension, arm flexion, arm extension, ankle flexion, and wrist extension. These results suggest that virtual reality sports applications could positively impact the development of strength parameters in children (Aykora et al., 2019).

The benefits of VR technology in enhancing cardiovascular health behaviors manifest in various dimensions. Regarding nutrition, interactive VR simulations can help users learn and practice healthy eating habits. In smoking cessation programs, VR environments can play a significant role by reducing cravings and supporting the quitting process. To promote physical activity, VR games make exercising fun, increase motivation, and improve activity levels. In combating sedentary lifestyles, VR exercises and activities can reduce sedentary time and encourage a more active lifestyle. In terms of stress reduction and self-esteem, VR environments can provide calming landscapes and a sense of achievement, thereby lowering stress levels and boosting self-esteem. This study aims to demonstrate that VR technology can be utilized as a multifaceted tool to improve cardiovascular health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Actively attending school where the research is conducted, Being a 6th-grade student, Willing to voluntarily participate in the research, Having written parental consent to participate in the research.

Exclusion Criteria:

* Interrupting the active education process during the research due to health problems or similar reasons, Changing schools, Having a chronic illness.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Data Collection Form | 5 weeks
  This form includes questions about the student's age, gender, height, weight, parental education level, family income level, the presence of a family member or close relative who has had a heart attack, and the presence of a family member or close relative using blood pressure medication.
Cardiovascular Health Behavior Scale for Children | 5 weeks
  The Cardiovascular Health Behavior Scale for Children was developed by Çelik and Bektaş to evaluate behaviors affecting children's cardiovascular health in a current and accurate manner (Çelik & Bektaş, 2020). The scale consists of subdimensions including nutrition, exercise, sedentary lifestyle, smoking, self-love, and stress.
  It measures cardiovascular health behavior levels with items such as "I eat chocolate, candy, or biscuits when I feel hungry, even if it's not mealtime," "I prefer to spend my free time doing sports," "I watch TV for more than 2 hours a day," "I feel uncomfortable when someone smokes near me," "I like my appearance," and "I worry about my schoolwork."
  The scale includes a total of 28 items scored on a 4-point Likert scale ranging from 1 (Always) to 4 (Never). While scoring, 15 items (1, 2, 3, 4, 5, 6, 7, 13, 14, 15, 16, 25, 26, 27, 28) are reverse-coded. Scores on the scale range from 28 to 112, with higher scores indicating a higher level of negative behavio

SECONDARY OUTCOMES:
Cardiovascular Health Behavior Scale for Children | 5 weeks
  The Cardiovascular Health Behavior Scale for Children was developed by Çelik and Bektaş to evaluate behaviors affecting children's cardiovascular health in a current and accurate manner (Çelik & Bektaş, 2020). The scale consists of subdimensions including nutrition, exercise, sedentary lifestyle, smoking, self-love, and stress.
  It measures cardiovascular health behavior levels with items such as "I eat chocolate, candy, or biscuits when I feel hungry, even if it's not mealtime," "I prefer to spend my free time doing sports," "I watch TV for more than 2 hours a day," "I feel uncomfortable when someone smokes near me," "I like my appearance," and "I worry about my schoolwork."
  The scale includes a total of 28 items scored on a 4-point Likert scale ranging from 1 (Always) to 4 (Never). While scoring, 15 items (1, 2, 3, 4, 5, 6, 7, 13, 14, 15, 16, 25, 26, 27, 28) are reverse-coded. Scores on the scale range from 28 to 112, with higher scores indicating a higher level of negative behavio

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Mehmet Çekiç Middle School, Ankara, Ankara
  - Sibel-İsmet Çatık Middle School, Ankara, Ankara

IPD SHARING:
Plan to Share IPD: No